CLINICAL TRIAL: NCT05020925
Title: A Phase I/II, Open-label, Multi-center Trial to Investigate the Efficacy and Safety of SHR-1701 in Combination With Famitinib in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: SHR-1701 in Combination With Famitinib in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-203-NPC
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; SHR-1701; Famitinib
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — SHR-1701; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 plus Famitinib (Experimental): SHR-1701+Famitinib for R/M NPC failure after platinum-based chemotherapy and anti PD-1/PD-L1 antibody therapy
  Interventions: Drug: SHR-1701; Drug: Famitinib

INTERVENTIONS:
Drug: SHR-1701 — Intravenous (IV) on Day 1 of each cycle
  Other Names: SHR-1701 Injection
Drug: Famitinib — Famitinib, po, qd
  Other Names: SHR-1020

SUMMARY:
This is an open label, multi-center, phase I/II study to evaluate the efficacy and safety of SHR-1701 in combination with famitinib in subjects with recurrent/metastatic nasopharyngeal carcinoma(R/M NPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Recurrent/Metastatic Nasopharyngeal Carcinoma
* Subjects failure after platinum-based chemotherapy and anti-PD-1/PD-L1 antibody therapy;
* Able and willing to provide signed informed consent form, and able to comply with all procedures.
* Life expectancy >= 12 weeks as judged by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry.
* Disease must be measurable with at least 1 uni dimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Adequate hematological, hepatic and renal function as defined in the protocol Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Anticancer treatment within 28 days before the first dose of study drug.
* Major surgery within 28 days before start of trial treatment.
* Systemic therapy with immunosuppressive agents within 7 days prior to the first dose of study drug; or use any investigational drug within 28 days before the start of trial treatment.
* With any active autoimmune disease or history of autoimmune disease.
* With active central nervous system (CNS) metastases causing clinical symptoms or requiring therapeutic intervention.
* History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immunedeficient disease, or any active systemic viral infection requiring therapy.
* Previous malignant disease (other than the target malignancy to be investigated in the trial) within the last 2 years. Subjects with history of cervical carcinoma in situ, superficial or non-invasive bladder cancer or basal cell or squamous cell cancer in situ previously treated with curative intent are NOT excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
ORR | up to approximately 2 years (anticipated)
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
DoR | up to approximately 2 years (anticipated)
  Duration of Response per RECIST 1.1
DCR | up to approximately 2 years (anticipated)
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1.
PFS | up to approximately 2 years (anticipated)
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
OS | up to approximately 2 years (anticipated)
  Overall Survival is defined as the time from registration to death due to any cause, or censored at date last known alive. OS will be measured by the Method of Kaplan and Meier.
AEs | up to approximately 2 years (anticipated)
  Number of participants with adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Guangzhou Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No